CLINICAL TRIAL: NCT03357809
Title: Monocentric Study Evaluating the Efficiency and Safety of Anti-reflux Mucosectomy ARMS for the Gastro-Esophageal Reflux Disease
Brief Title: Endoscopic Resection in Gastro-Esophageal Reflux Disease
Acronym: RESECT-RGO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lake of efficiency and poor tolerance of endoscopic technique
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Arthur Laquiere, Principal investigator, Hospital St. Joseph, Marseille, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01591-50
Record Dates: First submitted 2017-10-13; First posted 2017-11-30 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: GERD; Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic treatment (Experimental): ENDOSCOPIC MUCOSAL RESECTION AT DAY 1
  Interventions: Procedure: Endoscopic mucosal resection

INTERVENTIONS:
Procedure: Endoscopic mucosal resection — Mucosectomy performed at day 1. Endoscopic mucosal resection (EMR) and or endoscopic submucosal dissection (ESD), is at least 3 cm long. The mucosal resection is carried out along the side of the small curvature of the stomach, in order to preserve a valve of the cardia at the level of the large curvature of the stomach.
  A coloured solution is injected into the submucosa following markers. The correct submucosal injection is confirmed by the lifting of the mucosal surface. A submucosal dissection is carried out using the dual knife. The mucosectomy is repeatedly performed until the mucosal zone is completely resected. The choice of the resection technique will depend on the anatomy of the patient.

SUMMARY:
Currently patients with gastroesophageal reflux disease (GERD) are treated with proton pump inhibitors (PPIs). This long-term PPI treatment would likely increase the risk of pulmonary and digestive infections and would not prevent evolution to adenocarcinoma of Barrett's Esophagus. Surgical fundoplication is generally recommended when symptoms are poorly controlled with PPIs and considered as standard treatment despite celioscopy risk. A variety of endoscopic techniques for the treatment of GERD has been proposed to obtain non-surgical control. These endoscopic techniques aim to bring the tissues closer to the Œsogastric (JOG) junction. But a low response rate has been demonstrated with these techniques.

H. Inoue (inventor of the anti-reflux mucosectomy 20 years ago) and his team postulated that the reflux symptoms would be reduced by creating a relative restriction of gastric cardia. The healing of the mucosectomy zone led to restriction of gastric cardia. This observation suggested that ARMS could represent an effective anti-reflux procedure with the advantage that no prostheses would be left in situ.

Few studies have evaluated this new endoscopic technique. The purpose of this study is to evaluate the feasibility and safety of gastric mucosectomy for patients with GERD resistant to medical treatment or requiring long-term maintenance medical treatment.

DETAILED DESCRIPTION:
This is a monocentric prospective therapeutic study. Patients will be recruited in hepato-gastroenterology department of Saint Joseph Hospital (Marseille). A first clinical, endoscopic and PH impedance evaluation will be made. Mucosectomy will be scheduled depending on the results of the review.

The patients will be followed for 2 years with esophageal and gastric PH-impedance monitoring at 6 months and 24 months. Health related quality of life questionnaires will be completed before ARMS, 6 and 24 months after mucosectomy.

The characteristics of the patients will be compared to evaluate the % of responders and non-responders

ELIGIBILITY:
Inclusion Criteria:

* Patient with GERD resistant to medical treatment, or requiring daily long-term medical treatment

Exclusion Criteria:

* Contraindications to the realization of a upper GI endoscopy
* Achalasia or other esophageal motor disorders
* Voluminous hiatal hernia Haemorrhagic, haemostasis or coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-04-10 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients no longer requiring medical treatment at 6 months | 6 months
  Suggest that endoscopic treatment would allow the cessation of medical treatment in 50% of cases Rate of patients no longer requiring medical treatment at 6 months

SECONDARY OUTCOMES:
Improvement in quality of life | 6 months
  Percentage of improvement in quality of life measured by the score obtained in the GERD-HRQL questionnaire evaluating the impact of GERD on quality of life.
Improvement of gastric PH | 6 months
  Improvement of gastric PH metric dosages.
Evaluation for morbidity | 30 days
  Rate of all observed complications in per and post immediate procedure (up to 30 minutes). The delayed morbidity of the procedure for the study will be defined by the rate of complications occurring after the examination and up to 30 days. Specially, the following events will be studied: digestive hemorrhage and digestive perforation

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Laquière, MD, Principal Investigator — French Society of Digestive Endoscopy
Locations (1):
- LAQUIERE, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galmiche JP, Hatlebakk J, Attwood S, Ell C, Fiocca R, Eklund S, Langstrom G, Lind T, Lundell L; LOTUS Trial Collaborators. Laparoscopic antireflux surgery vs esomeprazole treatment for chronic GERD: the LOTUS randomized clinical trial. JAMA. 2011 May 18;305(19):1969-77. doi: 10.1001/jama.2011.626. PMID 21586712
- [Result] Cicala M, Emerenziani S, Guarino MP, Ribolsi M. Proton pump inhibitor resistance, the real challenge in gastro-esophageal reflux disease. World J Gastroenterol. 2013 Oct 21;19(39):6529-35. doi: 10.3748/wjg.v19.i39.6529. PMID 24151377
- [Result] Kellokumpu I, Voutilainen M, Haglund C, Farkkila M, Roberts PJ, Kautiainen H. Quality of life following laparoscopic Nissen fundoplication: assessing short-term and long-term outcomes. World J Gastroenterol. 2013 Jun 28;19(24):3810-8. doi: 10.3748/wjg.v19.i24.3810. PMID 23840119
- [Result] Marret H, Pierre F, Chapron C, Perrotin F, Body G, Lansac J. [Complications of laparoscopy caused by trocars. Preliminary study from the national registry of the French Society of Gynecologic Endoscopy]. J Gynecol Obstet Biol Reprod (Paris). 1997;26(4):405-12. French. PMID 9265066
- [Result] Rickenbacher N, Kotter T, Kochen MM, Scherer M, Blozik E. Fundoplication versus medical management of gastroesophageal reflux disease: systematic review and meta-analysis. Surg Endosc. 2014 Jan;28(1):143-55. doi: 10.1007/s00464-013-3140-z. Epub 2013 Sep 10. PMID 24018760
- [Result] Mahmood Z, Byrne PJ, McMahon BP, Murphy EM, Arfin Q, Ravi N, Weir DG, Reynolds JV. Comparison of transesophageal endoscopic plication (TEP) with laparoscopic Nissen fundoplication (LNF) in the treatment of uncomplicated reflux disease. Am J Gastroenterol. 2006 Mar;101(3):431-6. doi: 10.1111/j.1572-0241.2006.00534.x. PMID 16542276
- [Result] Triadafilopoulos G. Stretta: a valuable endoscopic treatment modality for gastroesophageal reflux disease. World J Gastroenterol. 2014 Jun 28;20(24):7730-8. doi: 10.3748/wjg.v20.i24.7730. PMID 24976710
- [Result] Feretis C, Benakis P, Dimopoulos C, Dailianas A, Filalithis P, Stamou KM, Manouras A, Apostolidis N. Endoscopic implantation of Plexiglas (PMMA) microspheres for the treatment of GERD. Gastrointest Endosc. 2001 Apr;53(4):423-6. doi: 10.1067/mge.2001.113912. PMID 11275880
- [Result] Cicala M, Gabbrielli A, Emerenziani S, Guarino MP, Ribolsi M, Caviglia R, Costamagna G. Effect of endoscopic augmentation of the lower oesophageal sphincter (Gatekeeper reflux repair system) on intraoesophageal dynamic characteristics of acid reflux. Gut. 2005 Feb;54(2):183-6. doi: 10.1136/gut.2004.040501. PMID 15647177
- [Result] Wong RF, Davis TV, Peterson KA. Complications involving the mediastinum after injection of Enteryx for GERD. Gastrointest Endosc. 2005 May;61(6):753-6. doi: 10.1016/s0016-5107(04)02645-8. No abstract available. PMID 15855987
- [Result] Chuttani R, Sud R, Sachdev G, Puri R, Kozarek R, Haber G, Pleskow D, Zaman M, Lembo A. A novel endoscopic full-thickness plicator for the treatment of GERD: A pilot study. Gastrointest Endosc. 2003 Nov;58(5):770-6. doi: 10.1016/s0016-5107(03)02027-3. PMID 14595322
- [Result] Cadiere GB, Buset M, Muls V, Rajan A, Rosch T, Eckardt AJ, Weerts J, Bastens B, Costamagna G, Marchese M, Louis H, Mana F, Sermon F, Gawlicka AK, Daniel MA, Deviere J. Antireflux transoral incisionless fundoplication using EsophyX: 12-month results of a prospective multicenter study. World J Surg. 2008 Aug;32(8):1676-88. doi: 10.1007/s00268-008-9594-9. PMID 18443855
- [Result] Satodate H, Inoue H, Yoshida T, Usui S, Iwashita M, Fukami N, Shiokawa A, Kudo SE. Circumferential EMR of carcinoma arising in Barrett's esophagus: case report. Gastrointest Endosc. 2003 Aug;58(2):288-92. doi: 10.1067/mge.2003.361. No abstract available. PMID 12872107
- [Result] Inoue H, Ito H, Ikeda H, Sato C, Sato H, Phalanusitthepha C, Hayee B, Eleftheriadis N, Kudo SE. Anti-reflux mucosectomy for gastroesophageal reflux disease in the absence of hiatus hernia: a pilot study. Ann Gastroenterol. 2014;27(4):346-351. PMID 25330784
- [Result] Velanovich V, Vallance SR, Gusz JR, Tapia FV, Harkabus MA. Quality of life scale for gastroesophageal reflux disease. J Am Coll Surg. 1996 Sep;183(3):217-24. PMID 8784314
- [Derived] Laquiere A, Trottier-Tellier F, Urena-Campos R, Lienne P, Lecomte L, Katsogiannou M, Penaranda G, Boustiere C. Evaluation of Antireflux Mucosectomy for Severe Gastroesophageal Reflux Disease: Medium-Term Results of a Pilot Study. Gastroenterol Res Pract. 2022 Feb 21;2022:1606944. doi: 10.1155/2022/1606944. eCollection 2022. PMID 35237316